CLINICAL TRIAL: NCT00579423
Title: A Pilot Multivalent Conjugate Vaccine Trial for Patients With Biochemically Relapsed Prostate Cancer
Brief Title: Multivalent Conjugate Vaccine Trial for Patients With Biochem. Relapsed Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Capcure (Unknown)
Responsible Party: Susan Slovin MD, PhD, Memorial Sloan-Kettering Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-064; NCT00016120 (obsolete NCT alias)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Prostate; Cancer
Keywords: prostate; cancer; vaccine
MeSH Terms: conditions — Neoplasms | interventions — saponin QA-21V1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccine (Experimental): Patients will be treated with specified doses of each carbohydrate or peptide constituent as has been determined. QS21 will be administrated at the standard dose of 100ug.
  Interventions: Biological: QS21

INTERVENTIONS:
Biological: QS21 — * Treatment schedule and dose: Thirty patients will be treated with specified doses of each carbohydrate or peptide constituent as has been determined. QS21 will be administered at the standard dose of 100 ug.
  * Sites: The vaccine conjugate will be administered subcutaneously on a rotating basis to random sites on the upper arms and upper legs.
  * Dose modifications: If a patient experiences a Grade III or greater local or Grade II or greater systemic toxicity at any time a decrease by 50% in all components of future vaccinations will be administered for that patient. Any evidence of autoimmunity, however, will result in a cessation of immunization in that patient.

SUMMARY:
This is a pilot trial designed to assess safety and immunogenicity of a multivalent conjugate vaccine for use in patients with biochemically relapsed prostate cancer.

DETAILED DESCRIPTION:
This is a pilot trial designed to assess safety and immunogenicity of a multivalent conjugate vaccine for use in patients with biochemically relapsed prostate cancer. This trial is based on the results of eight dose-seeking phase I monovalent glycoprotein and carbohydrate conjugate vaccine trials in a patient population with minimal tumor burden despite a rising biomarker, PSA, who have failed primary therapy such as surgery or radiation. We know that a rising PSA is indicative of micrometastatic disease - a state to which the immune system may maximally respond. Based on these trials, we have identified three glycolipid antigens, Globo H, Lewisy and GM2 and three mucin antigens, glycosylated MUC-1, Tn(c), and TF(c) for inclusion into a multivalent trial. As a result of these vaccinations, most patients generated specific high titer IgM and IgG antibodies against the respective antigen-KLH conjugates. Our previous work has shown the monovalent vaccines to be safe with local erythema and edema but minimal systemic toxicities. Our data from approximately 160 men who participated in our earlier monovalent vaccine trials against the aforementioned antigens have shown that a treatment effect in the form of a decline in PSA log slopes compared with pretreatment values could be seen in patients with minimal tumor burden. The multivalent vaccine will consist of the lowest dose of synthetic glycoprotein and carbohydrate antigens shown to elicit high titer IgM and IgG antibodies in patients with biochemically relapsed prostate cancer. A phase III double blind randomized trial with two hundred forty patients is planned based on the safety and immunogenicity data accrued from this pilot trial.

The primary endpoints of this study will be the safety of the vaccine and the humoral response to each of the antigens. The secondary endpoint will be to evaluate post-therapy changes in PSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer that is histologically confirmed.
* Patients must show biochemical progression after primary therapy, including surgery or radiation (with or without neo-adjuvant androgen ablation). This detection of PSA following treatment must occur within two years.
* Patients who have had intermittent hormonal treatment, following primary therapy, who have non-castrate levels of testosterone (>50 ng/ml) are eligible. Hormonal status will be recorded on the basis of serum testosterone levels.
* Karnofsky performance status >60%.
* Patients must have adequate organ function as defined by:

  1. WBC > or = to 3500/mm3, platelet count > or = to 100,000 mm3.
  2. Bilirubin <2.0 mg/100 ml or SGOT <3.0 X's the upper limit of normal.
  3. Creatinine < or = to 2.0 mg/100 ml or creatinine clearance > or = to 40 cc/min.
* Patients must have recovered from the toxicity of any prior therapy, and not received chemotherapy or radiation therapy for at least 4 weeks prior to entry into the trial.
* No history of an active secondary malignancy within the prior five years except for nonmelanoma skin cancer. Patients with history of melanoma in situ will be permitted since these lesions behave in a manner similar to compound nevi.
* Patients must be at least 18 years of age.
* Patients must sign informed consent.

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III/IV), or severe debilitating pulmonary disease.
* Radiographic evidence of metastatic disease.
* An infection requiring antibiotic treatment.
* Narcotic dependent pain.
* Anticipated survival of less than 6 months.
* Positive stool guaiac excluding hemorrhoids or history of documented radiation induced proctitis.
* Allergy to seafood.
* Prior vaccine therapy at outside institution except for phase I monovalent trial performed at MSKCC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-11; Primary Completion 2003-05 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Overall antitumor assessment performed during weeks 19 and 31. If no progression of disease continue on protocol. After week 31, will be monitored every 3 months with history, physical, performance status and bloodwork. Imaging studies every 6 mo. | 11/2000-12/2008

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org